CLINICAL TRIAL: NCT05207059
Title: Healthy Early Life Moments in Singapore
Acronym: HELMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Lien Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021/2247
Record Dates: First submitted 2021-12-22; First posted 2022-01-26 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Disease; Mental Health Wellness 1; Lifestyle Risk Reduction; Maternal Obesity
Keywords: Obesity; Mental health; Lifestyle intervention
MeSH Terms: conditions — Metabolic Diseases; Risk Reduction Behavior; Pregnancy in Obesity; Obesity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: HELMS is conceptualised as a single-arm implementation pilot trial, where lifestyle interventions are implemented in overweight or obese women from preconception to pregnancy and postpartum periods. We will follow both mother and child up to 18 months after delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): The intervention will comprise four modules, namely the HELMS Journey, HELMS Model, HELMS Lifestyle and HELMS Community. The HELMS Journey will provide anticipatory guidance for both HELMS and routine clinic visits. The HELMS Model will deliver the 4S ('Screening', 'Size', 'Supplementation' and 'Specific case management') care plan, detailed below. The HELMS Lifestyle will provide lifestyle support in terms of healthy eating through the 6P tool ('Portion', 'Proportion', 'Pleasure', 'Phase', Physicality', 'Psychology'), physical activity, sleep and mental well-being. Finally, the HELMS Connection will provide community support and improve engagement with the program.
  Interventions: Behavioral: HELMS Lifestyle Intervention

INTERVENTIONS:
Behavioral: HELMS Lifestyle Intervention — The HELMS life-course Interventions, namely 4S ('Screening', 'Size', 'Supplementation' and 'Specific case management'), are developed to deliver care throughout the journey from preconception to postpartum periods. Screening involves health and risk assessments through physical and biomarker measurements, as well as emotion and sleep evaluations for mother, and developmental assessment for children. Body Size management encompasses education on weight status awareness and mother-child health implications, both mother-child weight tracking, healthy eating and physical activity guidance. Supplementation includes multi-micronutrient, vitamin D, calcium and/or Docosahexaenoic acid (DHA) supplements, which is phase-specific for mother, and vitamin D drops supplement for child. Specific case management comprises preconception sexual health and function management, pregnancy symptoms management, postpartum recovery management, infant growth monitoring and feeding management.

SUMMARY:
This study aims to assess whether an integrated continuum of care from the preconception period, across maternity until the first 18 months of life, can promote maternal metabolic and mental health, as well as offspring health, among overweight and obese women.

DETAILED DESCRIPTION:
Maternal Child Health (MCH) in Singapore is currently entering a new phase to address the twin challenges; a burgeoning (i) Metabolic and (ii) Mental Health Challenge for Singapore which have shown to have adverse effects on childbearing and child outcomes. To tackle these challenges, we are establishing a new Model-of-Care (MOC) with a life-course approach at KK Women's and Children's Hospital (KKH) through the Healthy Early Life Moments in Singapore (HELMS) cohort. Over the course of five years, HELMS will enroll 500 overweight or obese women aged 21-40 years planning for pregnancy, with an estimated 170 completing their pregnancies where they will be followed for another 18 months as a mother-child dyad.

HELMS leverages on building a healthy mental model of life-course events through preconception to postpartum life. Components of intervention will focus on preconception-pregnancy-postpartum care and lifestyle guidance on diet, physical activity, emotion and sleep, complemented by health nudges to promote sustainable change. Various questionnaires and testing will be carried out at relevant time points. Biosamples including blood, cord blood and stool will be collected.

Through the application of HELMS, there is potential to improve metabolic and mental health, break vicious transgenerational cycles of obesity transmission and promote virtuous life cycles of health in the population.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 21-40 years
2. BMI 25-40 kg/m2
3. Intention to reside in Singapore for the next 4 years
4. Chinese, Malay, Indian or any combination of these 3 ethnic groups
5. Planning to conceive within 1 year
6. Able to understand English
7. Able to provide written, informed consent

Exclusion Criteria:

1. Currently pregnant
2. Known type 1 or type 2 diabetes
3. On any anticonvulsant medication in the past 1 month
4. On any oral steroid in the past 1 month (e.g. Prednisolone, Prednisone, Deltasone, Prelone, Methyl Prednisolone, Medrol, Hydrocortisone, Cortef, Dexamethasone, Decadron)
5. On any oral, implanted contraception or intrauterine contraceptive device (IUCD) in situ in the past 1 month
6. On any fertility medication (e.g. hormones injection, IVF treatments) other than Clomiphene/ Letrozole in the past 1 month
7. On HIV or Hepatitis B or C medication in the past 1 month.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | Up to 12 months
  Defined by positive urine pregnancy test, clinical diagnosis and/or ultrasound scan showing intrauterine gestation sac, in percentages
Maternal metabolic health | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Evaluated by metabolic syndrome criteria
Maternal mental health | Up to 26 months, between preconception, pregnancy and 4 months postpartum
  Measured by Edinburgh Postnatal Depression Scale, scored between 0 to 30, with a higher score being suggestive of depression

SECONDARY OUTCOMES:
Fecundability | Up to 12 months, between dates of last menstrual period at recruitment and before conception (for pregnant women) or last follow-up call (for non-pregnant women)
  Measured by time to pregnancy in total discrete cycles at risk of pregnancy
Female sexual function | Up to 3 months, between date of recruitment and 3 months preconception follow-up
  Measured by Female Sexual Function Index, with a higher score being suggestive of better sexual function
Pregnancy loss rate | Up to 42 weeks, between date of conception and date of delivery
  Based on ultrasound scan and medical records, in percentage
Live birth rates | Up to 42 weeks, between date of conception and date of delivery
  Based on ultrasound scan and medical records, in percentage
Maternal lipid levels | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Including total cholesterol, triglyceride, HDL-cholesterol, LDL-cholesterol, in mmol/L
Maternal glycaemic marker - plasma glucose | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by plasma glucose levels, in mmol/L
Maternal glycaemic marker - HbA1c | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by HbA1c, in percentage
Maternal glycaemic marker - C-peptide | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by C-peptide, in SI unit
Maternal glycaemic markers - Insulin | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by serum insulin, in SI unit
Maternal glucose tolerance status | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by Oral Glucose Tolerance Test (OGTT), in mmol/L
Maternal blood pressure | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by blood pressure device for systolic and diastolic pressures in mmHg
Maternal heart rate | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by blood pressure device or sensor in beats per minutes
Maternal body weight | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by weighing scale in kilograms
Maternal body weight status | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined by body mass index based on weight (kg) /height (m)2
Maternal body fat distribution | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from waist hip circumferences in centimeters
Maternal abdominal fat | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from waist hip circumferences in ratio
Maternal body composition | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from body fat analysis in percentages
Maternal body fat mass | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from body fat analysis in percentages
Maternal visceral fat | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from body fat analysis in volumes
Maternal body lean mass | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from body fat analysis in percentages
Maternal nutrient intake | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by food diary and/or food frequency questionnaire in SI units of respective nutrients
Maternal food intake | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by food diary and/or food frequency questionnaire in serving sizes
Maternal food intakes | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by food diary and/or food frequency questionnaire in grams
Maternal dietary pattern | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by food diary and/or food frequency questionnaire using factor loading analysis
Maternal food timing | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by food diary in time phase
Maternal eating episodes | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by food diary in eating frequency
Maternal dietary behaviour - 6P | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by 6P Questionnaire based on each factor in the questionnaire
Maternal dietary behaviour - TFEQ | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by Three Factor Eating Questionnaire, based on the scores from each category
Maternal micronutrient status | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Micronutrient panel from plasma or breastmilk such as 1-carbon metabolites, vitamin D and E, expressed in SI units of respective micronutrients
Maternal physical activity level - self assessment | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by International Physical Activity Questionnaire, with a higher score suggesting higher physical activity level
Maternal physical activity | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by accelerometer and/or digital sensor, in respective SI units
Maternal sedentary behaviour - self assessment | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by sedentary behaviour questionnaire, in hours and minutes per day, with longer duration suggestive of greater sedentary behaviour
Maternal sedentary behaviour | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by accelerometer and/or digital sensor, in respective SI units
Maternal sleep - PSQI | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by Pittsburgh Sleep Quality Index, scored from 0-21, with higher score suggestive of poor sleep quality
Maternal sleep | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by accelerometer and/or digital sensor, in respective SI units
Maternal emotional wellbeing | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by questionnaires
Maternal ocular health | Up to 21 months, from preconception until 36 weeks gestation
  Measured by retinal vessel characteristics (including vessel caliber, geometric assessment and vasoreactivity)
Maternal ocular health | Up to 21 months, from preconception until 36 weeks gestation
  Measured by retinal and choroidal characteristics using three-dimensional volumetric (OCT-A) imaging systems
Maternal personality trait | At preconception
  Measured by M5-50 questionnaire, with classification into respective personality types
Duration of gestation | Up to 42 weeks, between estimated date of conception from menstrual and ultrasound scan and date of delivery
  Defined as the length of pregnancy, in months and days
Number of participants with gestational diabetes | Up to 20 weeks, between 12 and 32 weeks gestation
  Determined by oral glucose tolerance test during pregnancy
Number of participants with hypertensive disorders of pregnancy | Up to 42 weeks, between date of conception and date of delivery
  Including pregnancy-induced hypertension and pre-eclampsia/eclampsia from questionnaire and/or retrieved from medical records
Mode of labour onset, course of delivery and delivery outcomes | Delivery
  From questionnaire and/or retrieved from medical records, reported in percentages
Maternal pain | Up to 5 months, between 32 weeks gestation and 6-8 weeks post-delivery
  Measured by pain questionnaire
Antenatal, perinatal and postnatal complications | Up to 50 weeks, between date of conception and up to 8 weeks postpartum
  From questionnaire and/or retrieved from medical records, reported in percentages
Neonatal complications and admission to neonatal care facilities | Up to 4 weeks, between date of delivery and 4 weeks post-delivery
  From questionnaire and/or retrieved from medical records, reported in percentages
Offspring body weight | Up to 18 months, from birth to infant age 18 months
  Weight measured in grams
Offspring body size at birth | At birth
  Adjusted for gestational age and sex, expressed in percentile
Offspring body length | Up to 18 months, from birth to infant age 18 months
  Measured in centimeters
Offspring head circumference | Up to 18 months, from birth to infant age 18 months
  Measured in centimeters
Intrauterine growth of foetus | Up to 30 weeks, between 7 weeks gestation and 37 weeks of gestation
  As assessed by antenatal serial ultrasound scans to determine head and abdominal circumference, femur length and estimated foetal weight
Offspring feeding | Up to 18 months, from birth to infant age 18 months
  Measured types of feeding using questionnaires
Offspring gut microbiome | Up to 18 months, from birth to infant age 18 months
  Measured from stool samples
Maternal gut microbiome | Up to 24 months, between preconception, pregnancy and 2 months postpartum
  Measured from stool samples
Influence of parental and offspring genotypes, body compositions, lifestyle and diet on the above primary and secondary outcomes | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by questionnaires, accelerometer, digital sensor and/or biomarkers
Acceptability and adherence levels | Up to 40 months, at preconception, pregnancy and 18 months postpartum
  From questionnaire, with higher score indicates higher acceptability and adherence
Satisfactory level of participants with the HELMS program | Up to 40 months, at preconception, pregnancy and 18 months postpartum
  From patient satisfaction questionnaire in a Likert scale, with a higher score suggesting greater satisfaction

OTHER OUTCOMES:
Health economics analysis of the HELMS program | Composite analysis between preconception visit which is up to 12 months before pregnancy and until infant age 18 months
  Cost benefit analysis from health expenses and diseases outcomes
Maternal general health and wellbeing | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From questionnaire, expressed in percentages
Offspring health and general wellbeing | Up to 18 months, from birth to infant age 18 months
  From questionnaire and/or medical records, expressed in percentages
Offspring metabolomic profile | Up to 18 months, from birth to infant age 18 months
  From cord blood, placenta, infant blood and/or skin biopsy
Offspring genomic profile | Up to 18 months, from birth to infant age 18 months
  From cord blood, placenta, infant blood and/or skin biopsy
Offspring epigenetic profile | Up to 18 months, from birth to infant age 18 months
  From cord blood, placenta, infant blood and/or skin biopsy
Offspring biochemical profile | Up to 18 months, from birth to infant age 18 months
  From cord blood, placenta, infant blood and/or skin biopsy
Offspring metabolic profile | Up to 18 months, from birth to infant age 18 months
  From cord blood, placenta, infant blood and/or skin biopsy
Offspring immunological profile | Up to 18 months, from birth to infant age 18 months
  From cord blood, placenta, infant blood and/or skin biopsy
Offspring molecular profile | Up to 18 months, from birth to infant age 18 months
  From cord blood, placenta, infant blood and/or skin biopsy
Maternal metabolomic profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood, urine and/or saliva samples
Maternal genomic profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood, urine and/or saliva samples
Maternal epigenetic profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood, urine and/or saliva samples
Maternal temperature | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by skin temperature sensor, in degree celsius
Maternal biochemical profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood, urine and/or saliva samples
Maternal metabolic profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood, urine and/or saliva samples
Maternal immunological profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood, urine and/or saliva samples
Maternal molecular profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood, urine and/or saliva samples
Paternal body weight | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Measured by weighing scale, in kilograms
Paternal body weight status | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined by body mass index based on weight (kg) /height (m)2
Paternal body fat distribution | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from waist hip circumferences in centimetres
Paternal abdominal fat | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from waist hip circumferences in ratio
Paternal body composition | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from body fat analysis in percentages
Paternal body fat mass | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from body fat analysis in percentages
Paternal body lean mass | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from body fat analysis in percentages
Paternal body visceral fat | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  Determined from body fat analysis in percentages
Paternal health and general well-being - self assessment | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From questionnaires
Paternal health and general well-being | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From digital sensor
Paternal immunological profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood and/or urine samples
Paternal biochemical profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood and/or urine samples
Paternal metabolic profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood and/or urine samples
Paternal molecular profile | Up to 40 months, between preconception, pregnancy and 18 months postpartum
  From blood and/or urine samples
Breast milk macronutrient profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
  From breast milk sample
Breast milk micronutrient profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
  From breast milk sample
Breast milk immune factor profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
  From breast milk sample
Breast milk epigenetic profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
  From breast milk sample
Breast milk biochemical profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
  From breast milk sample
Breast milk metabolic profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
  From breast milk sample
Breast milk microbiome profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
  From breast milk sample
Breast milk molecular profile (subsample) | Up to 1 year, between date of delivery and 1 year postpartum
  From breast milk sample
Maternal transcriptomics | Up to 36 months, between preconception, pregnancy and 1 year postpartum
  From blood and/or breast milk samples
Infant transcriptomics | Up to 36 months, between preconception, pregnancy and 1 year postpartum
  From blood

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Chan, MB BCh BaO MA FRCOG PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan JKY, Ku CW, Loy SL, Godfrey KM, Fan Y, Chua MC, Yap F. Effects of an integrated mobile health lifestyle intervention among overweight and obese women planning for pregnancy in Singapore: protocol for the single-arm healthy early life moments in Singapore (HELMS) study. BMJ Open. 2022 Dec 12;12(12):e061556. doi: 10.1136/bmjopen-2022-061556. PMID 36523242